CLINICAL TRIAL: NCT02110251
Title: Exercise Therapy With Risk Factor Management and Life Style Coaching After Vascular Intervention for Patients With Peripheral Arterial Disease With Critical Limb Ischemia or Tissue Loss. A Pilot Study
Brief Title: Exercise Therapy With Risk Factor Management and Life Style Coaching After Vascular Intervention for Patients With Peripheral Arterial Disease
Acronym: PEARL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with including patients
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Joep Teijink, prof. dr., Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEARL study
Record Dates: First submitted 2014-04-01; First posted 2014-04-10 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease, Rutherford 4 and 5 With Possibility to Improve Vascularization
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised exercise therapy (Experimental): Adequacy of initial therapy, Investigation degree of confusion and dementia, Preoperative preparation, Life-style coaching, Supervised Exercise therapy.
  Interventions: Behavioral: Supervised Exercise Therapy
- Walking advice (No Intervention): Standard care and a oral walking advice.

INTERVENTIONS:
Behavioral: Supervised Exercise Therapy
  Arms: Supervised exercise therapy

SUMMARY:
Patients with peripheral arterial disease with symptoms of critical ischemia or reduced tissue loss have a very high mortality and morbidity rate. So far, treatment strategies focused on the preservation of life and limb by an open surgical or endovascular revascularization, together with cardiovascular risk management and pain relief. Important modifiable factors related to mortality and morbidity are not covered in the current national and international guidelines. This study investigates the effects on mobility, mortality and quality of life with supplementation of the standard treatment of critical limb ischemia with supervised exercise therapy. Also a reduction of cardiovascular risk by intensive risk factor management and lifestyle coaching will be taken in to account. The supervised exercise therapy will take place under the supervision of a trained physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral arterial disease Rutherford stage 4 and 5, where it is possible to improve the vascularization of the affected leg with the help of an endovascular and / or open surgical vascular intervention.
* Patients with both legs are affected, but the most severe leg does not exceed stage 5.

Exclusion Criteria:

* Severe cardiopulmonary comorbidity (NYHA 4) and previous amputations of lower leg or thigh.
* Patients with limited amputation of the toes can participate.
* Insufficient understanding of the Dutch language.
* No physiotherapy insurance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mobility | 2 years
  Pain free walking distance WIQ ALDS

SECONDARY OUTCOMES:
Quality of life | 2 years
  RAND SF 36
Mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joep Teijink, prof. dr., Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (2):
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Medisch Centrum Alkmaar, Alkmaar